CLINICAL TRIAL: NCT01368198
Title: The Evaluation of Extended Tear Film Break Up Time (TFBUT) With an Ocular Emulsion
Brief Title: Evaluation of Extended Tear Film Break Up Time (TFBUT) With an Ocular Emulsion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Collaborators: Optometric Technology Group Ltd (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: ID11-10
Record Dates: First submitted 2011-05-06; First posted 2011-06-07 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-01

CONDITIONS: Dry Eye
Keywords: Ocular Emulsion; OPTIVE™ Lubricant; Tear Film Break Up Time
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ocular Emulsion (Active Comparator): An Ocular Emulsion
  Interventions: Other: Systane Balance Lubricating Eye Drops
- OPTIVE™ (Active Comparator): An OPTIVE™
  Interventions: Other: OPTIVE™

INTERVENTIONS:
Other: Systane Balance Lubricating Eye Drops — One instillation of the eye drop in each eye
  Other Names: Ocular Emulsion
  Arms: Ocular Emulsion
Other: OPTIVE™ — One instillation of the eye drop in each eye
  Other Names: Optive
  Arms: OPTIVE™

SUMMARY:
The primary objective of this investigation will be to quantify the increase in tear film break-up time (TFBUT) associated with the instillation of a single eyedrop of an Ocular Emulsion in dry eye sufferers.

DETAILED DESCRIPTION:
The secondary objective of this investigation will be to compare the tear film break up time measured with two different techniques.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must be 18 years of age or older;
2. The subject must have a best corrected visual acuity of 0.6 LogMAR (~6/24) or better in each eye
3. The subject must not have used any topical ocular drops for approximately 24 hours prior to the enrolment/screening visit
4. The subject must be classified as dry eye at enrolment/screening visit according to the following criteria:

   * Subjects' self-assessment of dry eye status (answer of at least "some of the time" to the question, "How often have your eyes felt dry enough to want to use eye drops?");
   * TFBUT measured with DET ≤ 5 seconds in at least one eye;
   * Grade 1 for meibomian gland expression in both eyes;
   * Evidence of missing meibomian glands in both eyes.

Exclusion Criteria:

1. History or evidence of ocular or intraocular surgery in either eye within the past six months.
2. History or evidence of serious ocular trauma in either eye within the past six months.
3. Current punctal occlusion of any type (e.g., collagen plugs, silicone plugs).
4. History or evidence of epithelial herpes simplex keratitis (dendritic keratitis); vaccinia; active or recent varicella viral disease of the cornea and/or conjunctiva; chronic bacterial disease of the cornea and/or conjunctiva and/or eyelids; mycobacterial infection of the eye; and/or fungal disease of the eye.
5. Use of any concomitant topical ocular medications during the study period.
6. Ocular conditions such as conjunctival infections, iritis, or any other ocular condition that may preclude the safe administration of either drop under investigation.
7. Participation in an investigational drug or device study within 30 days of entering this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2011-03; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Measurement of the tear film break-up time using DET sodium fluorescein strips. | Enrollment Test visit 1

SECONDARY OUTCOMES:
Measurement of the tear film break-up time in a non invasive manner using the Tearscope®. Measurement of the tear film break-up time in a non invasive manner using the Tearscope®. | Enrollment Test visit 2

CONTACTS AND LOCATIONS:
Locations (2):
- Contact Alcon Call Center for Trial Locations, Fort Worth, Texas, United States
- OTG Research & Consultancy, London, England, United Kingdom